CLINICAL TRIAL: NCT06021535
Title: Involvement of the Gut Microbiota and Its Metabolites in the Pathophysiology of Calcified Aortic Stenosis
Brief Title: Involvement of the Gut Microbiota in Calcified Aortic Stenosis
Acronym: Gut-CAS
Status: Not yet recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC Nr (2023-01173)
Record Dates: First submitted 2023-08-22; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Aortic Stenosis; Gastrointestinal Microbiome; Metabolomics
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, blood sample, aortic valve
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calcified Aortic Stenosis: Patients with calcified aortic valve or aortic stenosis will be enrolled Stool, blood samples and aortic valve of operated patients will be retrieved to evaluate the composition of the gut microbiota and its metabolites A follow up is planned for patients with no intervention on the aortic valve to assess the evolution of the aortic stenosis and the change in the gut microbiota.
  Interventions: Other: No intervention
- Control: Patients without calcified aortic valve will be enrolled Stool and blood samples will be retrieved to evaluate the composition of the gut microbiota and its metabolites No follow up is scheduled.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Calcific aortic stenosis (CAS) is a disease characterized by progressive calcification of the aortic valve, obstructing the passage of blood from the left ventricle into the general circulation. It is the most frequent cause of valve disease in the elderly. To date, no means of preventing the disease has been discovered, and the only treatment available is valve replacement during cardiac surgery, or percutaneous implantation of a valve prosthesis when the narrowing becomes severe and causes symptoms.

The intestinal flora or microbiota, the reservoir of all the microorganisms in the gut, is implicated in numerous diseases, particularly of the intestine. But to date, no study has established a link between CAS and microbiota. The intestinal microbiota acts through molecules produced by itself or the host and passing into the bloodstream. In the pathophysiology of CAS, the valve leaflets are breached and do not heal. These molecules can enter and have beneficial or deleterious effects, in particular promoting calcification of aortic valve cells.

Concrete objectives:

Improve understanding of calcific aortic stenosis in humans Study the composition of intestinal flora in patients with aortic stenosis and compare it with healthy subjects Study the molecules in the intestinal flora likely to be involved in the development of aortic stenosis in humans.

ELIGIBILITY:
Inclusion Criteria:

* Group of patients with CAS:
* Calcified aortic stenosis diagnosed on a cardiac ultrasound or CT not older than 3 months
* Severe aortic stenosis: surgical indication based on symptoms and ultrasound data (high gradient aortic stenosis : Vmax> 4m/s, mean gradient > 40mmHg, area < 1cm², low flow low-gradient CAS: left ventricular ejection fraction (LVEF) < 40%, Vmax< 4m/s, mean gradient < 40mmHg, area < 1cm², paradoxical low-gradient CAS: LVEF > 55%, Vmax< 4m/s, mean gradient < 40mmHg, area < 1cm²)
* Moderate CAS: 3m/s <Vmax< 4m/s, 20mmHg < mean gradient < 40mmHg
* Mild CAS: 2,6m/s < Vmax < 2.9m/s, mean gradient < 20mmHg
* Aortic sclerosis: calcified remodeling of the aortic valve visible on ultrasound or CT.

Control group - free of CAS:

- No calcified aortic stenosis verified on a cardiac ultrasound or CT not older than 3 months

Exclusion Criteria:

* Treatment interfering with the composition of the intestinal microbiota: local or systemic corticosteroids within the last 3 months, antibiotics within the last 3 months, antiretrovirals, bile acid chelators (questran and colesevelam), HIV-targeted antiretroviral therapies, selective serotonin reuptake inhibitor-type antidepressants
* Clinical criteria: history of cholecystectomy, documented chronic liver disease in the patient, failure to fast on the day of the blood test, inflammatory bowel disease
* Patients requiring emergency intervention (myocardial infarction, acute aortic or mitral insufficiency, cardiogenic shock).
* AS of rheumatic origin, infective endocarditis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study the investigators aim at enrolling patients with calcified aortic stenosis as well as a control group (patients without calcified aortic stenosis) and aim for an even distribution between female and male participants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Richness of the gut microbiota | The sample will be collected at the time of inclusion (with a margin of two additional days depending on the patient's ability to pass stools). The analysis will be performed at the end of the sample collection (an average of 2 years)
  The primary endpoint is the evaluation (16S ribosomal ribonucleic acid (rRNA) sequencing) of the species richness using alpha diversity parameters such as the Shannon and Simpson index and diversity between samples using beta diversity with Bray-Curtis dissimilarity approach. The investigators will then identify the bacteria with taxonomy analysis and statistical differences will be done using MaAsLin (Microbiome Multivariable Association with Linear Models) for patients with and without CAS.

SECONDARY OUTCOMES:
Comparison of the levels of the tryptophane metabolites of the gut microbiota in the blood, feces and the aortic valve between patients with and without CAS | The full analysis will be performed at the end of the sample collection. One intermediate analysis is scheduled when half of the samples are collected (one year and two years)
  The metabolites being studied include tryptophan metabolites (kynurenine pathway, serotonin pathway).
Comparison of the levels of the short chain fatty acids (SCFA) metabolites of the gut microbiota in the blood, feces and the aortic valve between patients with and without CAS | The full analysis will be performed at the end of the sample collection. One intermediate analysis is scheduled when half of the samples are collected (one year and two years)
  The metabolites being studied include SCFA (acetate, propionate and butyrate).
Comparison of the levels of the trimethylamine N oxide (TMAO) metabolites of the gut microbiota in the blood, feces and the aortic valve between patients with and without CAS | The full analysis will be performed at the end of the sample collection. One intermediate analysis is scheduled when half of the samples are collected (one year and two years)
  TMAO is derived from trimethylamine (TMA), itself generated by the action of the gut microbiota on dietary choline and phosphatidylcholine contained in red meat, eggs, dairy products and saltwater fish. TMAO and its derivatives (L Carnitine) are measured in blood, stool and valves.
Comparison of the levels of the bile acids metabolites of the gut microbiota in the blood, feces and the aortic valve between patients with and without CAS | The full analysis will be performed at the end of the sample collection. One intermediate analysis is scheduled when half of the samples are collected (one year and two years)
  The metabolites being studied include 4 bile acids and their derivatives (Cholic, Chenodeoxycholic, Deoxycholic and Lithocholic acid)
Diversity of bacteria families in men and women | The sample will be collected at the time of inclusion (with a margin of two additional days depending on the patient's ability to pass stools). The analysis will be performed at the end of the sample collection (an average of 2 years)
  Primary endpoint: The primary endpoint is the evaluation (16S rRNA sequencing) of the species richness using alpha diversity parameters such as the Shannon and Simpson index and diversity between samples using beta diversity with Bray-Curtis dissimilarity approach.
Prevalence of bacterial families or species in the microbiota of patients with CAS over the course of time and disease progression. | The sample will be collected at the time of inclusion (with a margin of two additional days depending on the patient's ability to pass stools). The analysis will be performed at the end of each year of follow up (an average of 2 years)
  Primary endpoint: The primary endpoint is the evaluation (16S rRNA sequencing) of the species richness using alpha diversity parameters such as the Shannon and Simpson index and diversity between samples using beta diversity with Bray-Curtis dissimilarity approach.
Prevalence of bacterial families or species in the microbiota of men versus women with CAS over the course of time and disease progression. | The sample will be collected at the time of inclusion (with a margin of two additional days depending on the patient's ability to pass stools). The analysis will be performed at the end of each year of follow up (an average of 2 years)
  Primary endpoint: The primary endpoint is the evaluation (16S rRNA sequencing) of the species richness using alpha diversity parameters such as the Shannon and Simpson index and diversity between samples using beta diversity with Bray-Curtis dissimilarity approach.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nguyen, MD, Principal Investigator — Insel Gruppe AG

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocyigit D, Tokgozoglu L, Gurses KM, Stahlman M, Boren J, Soyal MFT, Canpinar H, Guc D, Saglam Ayhan A, Hazirolan T, Ozer N. Association of dietary and gut microbiota-related metabolites with calcific aortic stenosis. Acta Cardiol. 2021 Jul;76(5):544-552. doi: 10.1080/00015385.2020.1853968. Epub 2020 Dec 18. PMID 33334254
- [Background] Liu Z, Li J, Liu H, Tang Y, Zhan Q, Lai W, Ao L, Meng X, Ren H, Xu D, Zeng Q. The intestinal microbiota associated with cardiac valve calcification differs from that of coronary artery disease. Atherosclerosis. 2019 May;284:121-128. doi: 10.1016/j.atherosclerosis.2018.11.038. Epub 2018 Dec 4. PMID 30897381
- [Background] Agus A, Planchais J, Sokol H. Gut Microbiota Regulation of Tryptophan Metabolism in Health and Disease. Cell Host Microbe. 2018 Jun 13;23(6):716-724. doi: 10.1016/j.chom.2018.05.003. PMID 29902437
- [Background] Shan Y, Pellikka PA. Aortic stenosis in women. Heart. 2020 Jul;106(13):970-976. doi: 10.1136/heartjnl-2019-315407. Epub 2020 Mar 22. PMID 32201373
- [Background] Morvan M, Arangalage D, Franck G, Perez F, Cattan-Levy L, Codogno I, Jacob-Lenet MP, Deschildre C, Choqueux C, Even G, Michel JB, Back M, Messika-Zeitoun D, Nicoletti A, Caligiuri G, Laschet J. Relationship of Iron Deposition to Calcium Deposition in Human Aortic Valve Leaflets. J Am Coll Cardiol. 2019 Mar 12;73(9):1043-1054. doi: 10.1016/j.jacc.2018.12.042. PMID 30846099
- [Background] Yilmaz B, Fuhrer T, Morgenthaler D, Krupka N, Wang D, Spari D, Candinas D, Misselwitz B, Beldi G, Sauer U, Macpherson AJ. Plasticity of the adult human small intestinal stoma microbiota. Cell Host Microbe. 2022 Dec 14;30(12):1773-1787.e6. doi: 10.1016/j.chom.2022.10.002. Epub 2022 Oct 31. PMID 36318918